CLINICAL TRIAL: NCT01847365
Title: Transcorneal Electrical Stimulation for the Treatment of Retinitis Pigmentosa - a Multicentre Safety Study of the Okustim® System
Brief Title: TES for the Treatment of RP
Acronym: TESOLAUK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TESOLAUK13
Record Dates: First submitted 2013-05-01; First posted 2013-05-06 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis Pigmentosa; Transcorneal electrical stimulation; Okustim
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Retinitis Pigmentosa (Experimental): Transcorneal electrical stimulation (TES) administered to one eye for 6 months, followed by monitoring period without treatment for 6 months.
  Interventions: Device: Transcorneal electrical stimulation

INTERVENTIONS:
Device: Transcorneal electrical stimulation — Transcorneal electrical stimulation will be delivered by the CE-marked Okustim device.

SUMMARY:
Retinitis pigmentosa (RP) is a progressive degenerative disease of the retina, which often leads to blindness. 1 in 4000 people in the UK are affected by RP yet there is no established therapy for treating or delaying its progression.

Transcorneal electrical stimulation (TES) has garnered attention as a possible therapeutic option for RP. Research has shown that TES improves retinal cell viability and visual function. An initial pilot study of TES on 24 participants with RP demonstrated that it was safe and improved vision.

This study aims to confirm the safety of the new CE-approved Okustim device and to further characterise the benefits of TES on a larger scale. 12 participants will be enrolled for 1 year across two sites in the UK - the Oxford Eye Hospital and London Moorfields Eye Hospital.

Recruited participants will undergo weekly TES of 1 eye for 30 minutes for a period of 6 months. This will be followed by a further 6 months of observation without stimulation giving a total participation time of 1 year. Participants will be assessed at 3, 6, 9 and 12 months after their initial baseline visit by clinical examination, investigations and questionnaires.

Participants should have a diagnosis of RP and be capable of giving consent. Participants, or a carer, should have sufficient motor skills to attach the device themselves. As this study seeks to ascertain the impact of TES on RP, participants with other eye diseases (e.g. diabetic retinopathy) cannot be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Male or Female, 18 or more years of age
* Diagnosis of retinitis pigmentosa (rod-cone dystrophy) made by an ophthalmologist
* Participants should have a visual acuity of ≥ 0.02 (Snellen Chart)
* Able (in the investigators opinion) and willing to comply with all study requirements
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study
* Participants, or a designated other, should have sufficient motor skills (assessed by the investigator) to apply the device independently

Exclusion Criteria:

* Female participants who are pregnant, lactating or planning pregnancy during the course of the study
* Diabetic Retinopathy
* Previous arterial or venous occlusion of the retina
* Previous retinal detachment
* Previous silicone oil tamponade
* Dry or exudative age-related macular degeneration
* Macular oedema
* All forms of glaucoma
* Any form of corneal degeneration that reduces visual acuity
* Neovascularisation of any origin
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study
* Forms of mental illness related to bipolar affective and schizoid-affective disorders, and all forms of dementia
* Simultaneous participation in another interventional study or history of interventions where effects may still persist

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 12 months
  Quantity and Character of Adverse Events Related to the Use of the Device

SECONDARY OUTCOMES:
Efficacy of Intervention | 12 months
  Ophthalmic examination, best corrected visual acuity, visual field assessment, microperimetry, optical coherence tomography, fundus photography

OTHER OUTCOMES:
Usability of the Device | 12 months
  Non-validated questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Robert E MacLaren, FRCOphth DPhil, Study Chair — University of Oxford, Oxford University Hospitals NHS Trust and Moorfields Eye Hospital NHS Foundation Trust; Susan M Downes, FRCOphth MD, Principal Investigator — Oxford University Hospitals NHS Trust and University of Oxford; Andrew R Webster, FRCOphth MD, Principal Investigator — UCL Institute of Ophthalmology and Moorfields Eye Hospital NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Oxford University Hospitals NHS Trust, Oxford, Oxfordshire
  - Moorfields Eye Hospital NHS Foundation Trust, London

REFERENCES:
- [Background] Jolly JK, Wagner SK, Moules J, Gekeler F, Webster AR, Downes SM, MacLaren RE. A Novel Method for Quantitative Serial Autofluorescence Analysis in Retinitis Pigmentosa Using Image Characteristics. Transl Vis Sci Technol. 2016 Dec 1;5(6):10. doi: 10.1167/tvst.5.6.10. eCollection 2016 Dec. PMID 27933220
- [Result] Wagner SK, Jolly JK, Pefkianaki M, Gekeler F, Webster AR, Downes SM, Maclaren RE. Transcorneal electrical stimulation for the treatment of retinitis pigmentosa: results from the TESOLAUK trial. BMJ Open Ophthalmol. 2017 Dec 14;2(1):e000096. doi: 10.1136/bmjophth-2017-000096. eCollection 2017. PMID 29354722
- See also: Oxford Eye Hospital — http://www.eye.ox.ac.uk